CLINICAL TRIAL: NCT04944732
Title: Follow up Evaluation of Diagnostic Criteria for Creutzfeldt Jakob Disease (WS / T 562-2017)
Brief Title: Evaluation of Diagnostic Criteria for Creutzfeldt Jakob Disease
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Centers for Disease Control and Prevention, China (Other Government)
Responsible Party: Sponsor
Other Study IDs: M2020331
Record Dates: First submitted 2021-06-27; First posted 2021-06-30 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Creutzfeldt Jakob Disease
MeSH Terms: conditions — Creutzfeldt-Jakob Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Creutzfeldt Jakob disease: Patients with Creutzfeldt Jakob disease
  Interventions: Diagnostic Test: laboratory examination, auxiliary examination, pathological results

INTERVENTIONS:
Diagnostic Test: laboratory examination, auxiliary examination, pathological results — Personal information (sex, age), medical history of present disease, past medical history, family history, symptoms and signs, supplementary examination items (including laboratory examination, impact examination)

SUMMARY:
Clinicians know little about Creutzfeldt Jakob disease, and they are not proficient in the diagnostic criteria of Creutzfeldt Jakob disease, so it is easy to misdiagnose or delay the diagnosis. As a rare central nervous system disease, it is necessary, feasible and practical to evaluate the diagnostic criteria of Creutzfeldt Jakob disease.

DETAILED DESCRIPTION:
To master the clinical application of the diagnosis of Creutzfeldt Jakob disease (WS / T 562-2017) and the problems in the implementation process; The rationality, practicability and operability of the diagnostic criteria were evaluated scientifically; Reduce the misdiagnosis rate; To provide clinical basis and suggestions for further improving the diagnostic criteria. Through consulting the literature of Creutzfeldt Jakob disease, the clinical manifestations, laboratory examination, auxiliary examination and pathological results of Creutzfeldt Jakob disease were analyzed and compared with the current diagnostic criteria; The clinical diagnosis and misdiagnosis of Creutzfeldt Jakob disease were analyzed; To train medical staff at all levels to apply the diagnostic criteria of Creutzfeldt Jakob disease, and to discuss the clinical cases of Creutzfeldt Jakob disease in many hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Creutzfeldt Jakob disease

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Creutzfeldt Jakob disease
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Clinical manifestations | 1 year
  Clinical manifestations of patients

CONTACTS AND LOCATIONS:
Overall Officials: Li Xiaogang, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No